CLINICAL TRIAL: NCT04671108
Title: Comparative Clinical Performance of 59% Hioxifilcon A Daily Disposable Contact Lenses vs. Marketed Daily Disposable Hydrogel Contact Lenses
Brief Title: Comparative Clinical Performance of 59% Hioxifilcon A Contact Lenses vs. Marketed Hydrogel Contact Lenses
Acronym: DDHyd
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vision Service Plan (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: VS-20-02
Record Dates: First submitted 2020-12-07; First posted 2020-12-17 (Actual); Last update posted 2021-07-23 (Actual); Status verified 2021-07

CONDITIONS: Refractive Error - Myopia Bilateral

STUDY DESIGN:
Intervention Model Description: Randomized cross-over with 1 week of lens wear with each contact lens type.
Who Masked: Care Provider
Masking Description: Clinician masking achieved by clinic coordinator dispensing lenses. Open label to participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Test to Moist (Experimental): 1 week of Test DD contact lenses followed by cross over to 1 week of 1-DAY ACUVUE® Moist contact lenses.
  Interventions: Device: Hioxifilcon A standard hydrogel contact lens with Hyaluronic Acid (HA)
- Moist to Test (Active Comparator): 1 week of 1-DAY ACUVUE® Moist contact lenses followed by cross over to 1 week of Test DD contact lenses.
  Interventions: Device: Hioxifilcon A standard hydrogel contact lens with Hyaluronic Acid (HA)

INTERVENTIONS:
Device: Hioxifilcon A standard hydrogel contact lens with Hyaluronic Acid (HA) — Daily disposable contact lens wear for 1 week

SUMMARY:
The study will compare the short-term clinical performance and wearer and practitioner acceptability of a new-to-market spherical daily disposable (DD) hydrogel soft contact lens to a currently marketed spherical DD hydrogel soft contact lens.

DETAILED DESCRIPTION:
This randomized clinical trial will compare the short-term clinical performance, and wearer acceptability of a new-to-market hioxifilcon A spherical daily DD contact lenses against marketed DD lenses in a short cross-over clinical trial.

The primary outcome variable for this study is overall subjective comfort.

ELIGIBILITY:
Inclusion Criteria:

* Currently wearing spherical DD contact lenses at least 5 days/week
* Vision correctable to 20/30 acuity in each eye with spherical DD contact lenses
* No ocular or systemic disease that contra-indicates soft contact lens wear

Exclusion Criteria:

* Participating in another clinical trial
* Vision not correctable to 20/30

Ages: 18 Years to 42 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2020-11-11 (Actual); Primary Completion 2020-12-18 (Actual); Study Completion 2020-12-18 (Actual)

PRIMARY OUTCOMES:
Overall subjective comfort | 1 week after contact lens wear
  Subjective comfort rating on a scale of 0 (Painful) to 10 (Can't feel the lenses)
Overall subjective comfort | 2 weeks after contact lens wear
  Subjective comfort rating on a scale of 0 (Painful) to 10 (Can't feel the lenses)

SECONDARY OUTCOMES:
End of day subjective comfort | Visit 2 and 3 - Approximately 1 and 2 weeks, respectively
  Subjective comfort rating on a scale of 0 (Painful) to 10 (Can't feel the lenses)
Subjective vision | Visit 2 and 3 - Approximately 1 and 2 weeks, respectively
  Subjective vision rating on a scale of 0 (Not at all sharp/clear) to 10 (Sharp/Clear)
Overall subjective lens preference | Visit 3 - After approximately 2 weeks of contact lens wear
  Forced choice subjective preference for either lens type (1-Day ACUVUE® MOIST or Test DD contact lens) or no preference. i.e. three options presented and participant selects one option.

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Ross Eyecare, Atlanta, Georgia
  - Professional VisionCare, Westerville, Ohio
  - Primary Eyecare Group, Brentwood, Tennessee

IPD SHARING:
Plan to Share IPD: No